CLINICAL TRIAL: NCT02419235
Title: The Effect of a Homoeopathic Complex (Amylenum Nitrosum 6CH, Crataegus Oxyacantha 6CH, Natrum Muriaticum 6CH and Scutellaria Lateriflora 6CH) on Blood Pressure in Refractory Hypertension
Brief Title: The Effect of a Homoeopathic Complex on Blood Pressure in Refractory Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr J. Pellow, University of Johannesburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NangamsoBavuma200907364
Record Dates: First submitted 2015-04-04; First posted 2015-04-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Essential Hypertension
Keywords: Refractory hypertension; Homoeopathy; Homoeopathic complex; Amylenum nitrosum 6cH; Crataegus oxyacantha 6cH; Natrum muriaticum 6cH; Scutellaria lateriflora 6cH
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20% Ethanol (Placebo Comparator): Ten drops of unmedicated 20% ethanol must be administered under the tongue, three times per day, thirty minutes before or after meals, for six weeks.
  Interventions: Other: 20% ethanol
- Homoeopathic complex (Experimental): Ten drops of 20% ethanol medicated with Amylenum nitrosum 6cH, Crataegus oxyacantha 6cH, Natrum muriaticum 6cH and Scutellaria lateriflora 6cH will be administered under the tongue, three times per day, thirty minutes before or after meals, for six weeks.
  Interventions: Other: Homoeopathic complex

INTERVENTIONS:
Other: 20% ethanol — Unmedicated 20% ethanol.
  Other Names: 20% alcohol
  Arms: 20% Ethanol
Other: Homoeopathic complex — 20% ethanol medicated with Amylenum nitrosum 6cH, Crataegus oxyacantha 6cH, Natrium muriaticum 6cH and Scutellaria lateriflora 6cH.
  Arms: Homoeopathic complex

SUMMARY:
Refractory hypertension is defined as failure to reach goal blood pressure control in patients who are adherent to full doses of the appropriate drug regime. Hypertension results in 7.6 million deaths annually and 92 million disability adjusted years worldwide, making it the number one attributable risk for death throughout the world. Conventional treatment involves lifestyle modification and antihypertensive drug therapy; however blood pressure can remain uncontrolled despite these treatment options. Previous studies have demonstrated a reduction in blood pressure in adults with essential hypertension with the use of various homoeopathic complexes. There has been no research done to date on the effect of the homoeopathic combination of Amylenum nitrosum 6cH, Crataegus oxyacantha 6cH, Natrum muriaticum 6cH and Scutellaria lateriflora 6cH in adults with refractory hypertension.

The aim of the study is to investigate the effect of a homoeopathic complex Amylenum nitrosum 6cH, Crataegus oxyacantha 6cH, Natrum muriaticum 6cH and Scutellaria lateriflora 6cH on blood pressure in adults with refractory hypertension, by means of blood pressure readings.

DETAILED DESCRIPTION:
This study is a six week, double-blind, placebo-controlled pilot study. Thirty participants, aged 35 to 60 years, who have been previously diagnosed by their healthcare provider with refractory hypertension, will be recruited by means of purposive sampling. Adverts will be placed at the University of Johannesburg (UJ) Doornfontein campus and the Soweto satellite clinic Nanga Vutshilo Community Centre.

Potential participants that respond to the advert will attend an initial consultation and will be requested to sign a Participant Information and Consent Form once they agree to participate in the study. The medical history and physical examination (including vital signs, fundoscopic exam, cardiovascular exam, respiratory exam and urinalysis) will be recorded on a Case Form. Blood pressure (BP) readings will be taken on each arm with a manual BP cuff, according to standard operating procedures, on the first three consecutive days to confirm inclusion into the study. Individuals with secondary organ damage from hypertension will be excluded from the study.

Those participants that qualify for the study will be placed into two groups. One group will receive a 50ml bottle of the homoeopathic complex and the other group a 50ml bottle of placebo. Participants will receive an Intake Diary, to be completed daily, recording compliance and any adverse symptoms or aggravations that may be experienced. Follow-up consultations will take place every 7 days and participants will be requested to bring with their medication bottles for further assessment of compliance; BP readings will be recorded on a data collection form. All participants will be given the Dietary Approaches to Stop Hypertension (DASH) eating plan at the end of the study to help control their hypertension. Additionally, participants will be given an information leaflet to give to their healthcare provider, detailing the study.

Data will be analysed using the non-parametric methods: inter-group analysis will be conducted using SPSS v18 with the Mann-Whitney U-test; intra-group analysis will be done using the Friedman and the Wilcoxon-Signed Ranks tests.

A possible outcome of this study is that the homoeopathic complex will have a normalizing effect on BP readings compared to placebo. Regardless of the outcome, this study will contribute to our knowledge on the use of homoeopathic complex remedies in the treatment and management of refractory hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female, between the ages of 35-60 years;
* have a systolic blood pressure between 140 mmHg-160 mmHg;
* have a diastolic blood pressure between 90 mmHg-99 mmHg; and
* are on 3 or more conventional anti-hypertensive medications of different drug classes, one of which must be a diuretic.

Exclusion Criteria:

* Have a systolic blood pressure < 140 mmHg; > 160 mmHg;
* have a diastolic blood pressure < 90 mmHg; > 99 mmHg;
* are pregnant or lactating;
* are on any other herbal or homoeopathic medicine for the treatment of hypertension;
* have secondary organ damage from hypertension; and or
* suffer from chronic conditions such as severe cardiac disease, renal failure, malignant hypertension or diabetes mellitus.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Weekly blood pressure measurements using a Dura Shock Handheld Aneroid sphygmomanometer model DS55 | 6 weeks
  Blood pressure will be monitored in the left and right arm of each participant with a Dura Shock Handheld Aneroid sphygmomanometer model DS55, which will be correctly calibrated. An obese BP cuff will be used for overweight participants to ensure reliable results. Blood pressure measurements will be conducted according to standard operating procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Pellow, M.TechHom, Study Director — University of Johannesburg
Locations (1):
- University of Johannesburg, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No